CLINICAL TRIAL: NCT01650363
Title: Effect of Complementary and Alternative Medical Methods on the Post Operative Recovery Following Cardio-thoracic Surgery- a Pragmatic, Randomized,Single Blinded, Placebo Controlled Study
Brief Title: CAM in Post Surgical Management in Cardiothoracic Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Menachem Oberbaum, MD, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTSURG
Record Dates: First submitted 2012-07-16; First posted 2012-07-26 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Patients Undergoing Open Heart Surgery; Patients Undergoing Lung Surgery
Keywords: Complementary and alternative medicine; Post operative recovery; Cardio- thoracic surgery
MeSH Terms: interventions — Acupuncture Therapy; Homeopathy; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture, homeopathy, osteopathy and reflexology (Active Comparator): patients will receive combinations of acupuncture, homeopathy, osteopathy and reflexology
  Interventions: Other: Acupuncture, homeopathy, osteopathy- and reflexology
- homeopathic placebo medication (Placebo Comparator)
  Interventions: Drug: Homeopathic placebo medication

INTERVENTIONS:
Other: Acupuncture, homeopathy, osteopathy- and reflexology — a combination of the above mentioned treatments
  Arms: Acupuncture, homeopathy, osteopathy and reflexology
Drug: Homeopathic placebo medication — 2-3 mm small spheric suger pils
  Arms: homeopathic placebo medication

SUMMARY:
This is a randomized controlled clinical trial in which the combination of 4 different CAM modalities (Complementary & Alternative Medicine) will be applied during the postoperative period to patients undergoing open heart- or lung surgery and expected to be hospitalized for more than 5 days.

Elective and Urgent surgical patients will be randomly assigned to a treatment - and to a control group. The treatment group will be treated with a combination of 4 different CAM modalities (Homeopathy, Osteopathy, and Acupuncture & Reflexology) . The control group will be treated with Homeopathic placebo medication.

The main Outcome measurement in the study will be the Quality of recovery 40 questionnaire (QoR- 40) that will be filled out on postoperative days: 3, 5, and 7 respectively. Secondary outcome measurements will be Blood &Saliva Cortisol levels, DHES levels in the blood as surrogates of stress, IL-2 levels as measures of the immune system. Further parameters to be measured include: LOS (length of stay), Level of Pain, mobility, level of satisfaction, GI symptoms (nausea, first bowel movement), post-operative complications& side effects.

All patients participating in the trial will sign an informed consent form . The trial is expected to be conducted over a period of 12 months. Prior to the trial a pilot study will be conducted on a group of 30 patients in order to determine the needed sample size for the trial.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Patients planned to undergo a surgical procedure which will require an estimated hospitalisation of at least 5 days
* Patients speaking Hebrew or English
* Informed Consent signature

Exclusion Criteria:

* patients unable to comply with the study protocol
* Participation in another clinical trial
* Thrombocytopenia (< 15.000 for acupuncture treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Improvement of Quality of Recovery questionnaire-40 (QoR-40) | days 3,5 and 7
  Quality of Recovery questionnaire is a tool which is used primarily to assess the patient's recovery and state of health following surgery.

SECONDARY OUTCOMES:
Stress levels | Study entry, 2nd and 3rd day following the treatment initiation.
  Level of stress will be determined by Dehydroepiandrosterone (DHES) & Cortisol levels in blood and, saliva.
Immune System Function | 2nd and 4th day after treatment initiation
  - the function of the immune system will be evaluated by measuring IL-2 level on the second and fourth day
Length of Stay | patients will be followed for the duration of the hospital stay, an expected average of 4 weeks
  Hospitalization duration will be calculated from the first postoperative day. Readiness for discharge will be assessed based on the following measures: Bowel movements and lack of urinary retention yes/no; Ability to dress oneself and move freely; opiate requirement yes/no. Surgical complications requiring further hospitalization yes/no.
  Readiness for discharge will be based on a 'YES " for the first 2 measures and a "no" ON THE LAST 2 MEASURES.
First postoperative passage of flatus and first bowel movement. | the time to the first passage of flatus and bowel movements, an expected average of 3 days
GI Symptoms | patients will be evaluated for GI symptoms until discharge (expected average 4 weeks)
  Nausea levels and frequency of vomiting
Food intake | participants will be evaluated for the ingestion of the first solid meal (average: 4 days)
  Duration from surgery to first solid meal
Analgesia Protocol | daily intake of anlagesic medications will be evaluated each evening throughout the study period (mean expected: 4 weeks)
  Analgesics use
Pain level estimation | first 3 days and day 6
  Pain estimation will be based on the NRS scale. The patient will be asked to rate the highest level of pain experienced during the last 24 hrs.
Fatigue | Daily at 3rd, 4th and 5th post operative days 3,4 and 5
  0- 10 scale (0=no fatigue; 10 maximal fatigue)
Ambulation | each day participants will be evaluated for ambulation (expected mean: 1 week)
  As ambulant will a patient regarded if he will be able to walk 5 minutes without help
Patient Satisfaction | at discharge from hospital; expected mean: 4 weeks
  Patient satisfaction questionnaire
Hospitalization costs | At hospital discharge (mean expected: 4 weeks)
Postoperative complications | Every day, to be evaluated each evening throughout the hospital stay (mean expected: 4 weeks)
Side-effects | every day; to be evaluated each evening throughout the study period (mean expected: 4 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Menachem Oberbaum, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Dptm. Cardio-Thoracic Surgery, Shaare Zedek medical Center, Jerusalem, Israel